CLINICAL TRIAL: NCT05522023
Title: The Effect of Aromatic Solution Applied After Percutaneous Nephrolithotomy Surgery on Sore Throat, Thirst and Nausea-Vomiting
Brief Title: Effects of Aromatic Solution Applied After Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Esma Gökçe, Principal Investigator (MSc), Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 466455
Record Dates: First submitted 2022-08-25; First posted 2022-08-30 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Surgery; Nurse's Role; Throat, Sore; Thirst; Nausea and Vomiting, Postoperative
Keywords: surgical nursing; complementary alternative medicine; non-pharmacological applications; post-operative care; aromatherapy; sore throat; thirst; nausea vomiting
MeSH Terms: conditions — Pharyngitis; Postoperative Nausea and Vomiting | interventions — Drinking Water

STUDY DESIGN:
Intervention Model Description: 3 group randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (group treated with aromatic solution) (Experimental): Informed consent form will be signed by the patients selected by randomization and a personal information form will be filled.
  Hour 0: The patients will be completely awakened from the anesthesia resting unit, their vital signs will be stable, they will be transferred to the clinic where they lie normally with a 15 glaskow scale, the bed head will be elevated 45 degrees and the risk of aspiration will be ruled out. After controlling the vital signs of the patient, sore throat and thirst with VAS and nausea and vomiting with the verbal descriptive scale VDS will be evaluated. After the data are collected, the aromatic solution will be shaken and applied to the oral cavity and throat as a spray 4 times. After the aromatic solution application is finished, the patients' sore throat, thirst and nausea and vomiting will be re-evaluated with the same forms.
  2., 4., 6. The same procedures will be repeated in the 8th and 8th hours.
  Interventions: Procedure: group treated with aromatic solution
- Placebo group (group treated with drinking water) (Placebo Comparator): Patients included in this group as a result of randomization will have to sign an informed consent form and fill out a personal information form.
  Hour 0: The patients will be completely awakened from the anesthesia resting unit, their vital signs will be stable, they will be transferred to the clinic where they sleep normally with a 15 glaskow scale, the bed head will be elevated 45 degrees and the risk of aspiration will be ruled out. Nausea and vomiting will be evaluated with a verbal descriptive scale. After the data are collected, drinking water will be applied to the oral cavity and throat in the form of a spray 4 times. After the drinking water application is finished, the patients' sore throat, thirst and nausea and vomiting will be re-evaluated with the same forms.
  2., 4., 6. The same procedures will be repeated in the 8th and 8th hours.
  Interventions: Procedure: group treated with drinking water
- Control Group (No Intervention): Patients in the control group were planned to be followed according to their clinical procedures. Since there were no procedures or interventions in the clinical procedures, it was decided to follow up only the patient, and the control group patients to be followed up at the same times with the same forms.
  Patients included in this group as a result of randomization will have to sign an informed consent form and fill out a personal information form. Hour 0: Patients will be transferred from the recovery unit to the clinic. After controlling the vital signs of the patient, sore throat and thirst with VAS and nausea and vomiting with a verbal descriptive scale will be evaluated. 2., 4., 6. The same procedures will be repeated in the 8th and 8th hours.

INTERVENTIONS:
Procedure: group treated with aromatic solution — The aromatic solution applied in the experimental group will be obtained by mixing lavender oil and ginger oil into cold drinking water. For this, lavender and ginger oil approved by the Ministry of Agriculture will be used. 3 drops of lavender oil and 3 drops of ginger oil will be mixed into each 100 ml of drinking water, and it will be applied by spraying 4 times in the oral cavity and throat by shaking to ensure homogeneous distribution before each use. The aromatic solution to be applied in the study will be applied with spray bottles with mouth caps and caps that will be specially provided for each patient.
  Arms: Experimental group (group treated with aromatic solution)
Procedure: group treated with drinking water — In the placebo group, drinking water will be sprayed 4 times in the oral cavity and throat of the patients after the surgery. The aromatic solution to be applied in the study will be applied with spray bottles with mouth caps and caps that will be specially provided for each patient.
  Arms: Placebo group (group treated with drinking water)

SUMMARY:
Today, surgical applications are used to solve many health problems. In order for the surgical intervention to take place, anesthesia applications are often required. Complications such as sore throat, thirst and nausea and vomiting may occur as a result of trauma, local irritation and inflammation of the airway mucosa during anesthesia and tracheal intubation. These complications are in the postoperative period; It may cause delayed oral fluid intake, prolonged dehydration, oral odour, and increased risk of aspiration, hematoma and wound dehiscence due to retching and vomiting, all of which may lead to delayed discharge and increased cost. Aromatherapy, one of the non-pharmacological applications, is frequently applied in reducing postoperative complications and its effectiveness is stated.

In this study, the aromatic solution applied after the surgery; It was planned to examine the effect on sore throat, thirst, nausea-vomiting. In addition, the multimodal synergistic effect of lavender oil and ginger oil used in the aromatic solution to be prepared will be utilized. As a result of this study, the effectiveness of the aromatic solution application to be applied to the patients in the postoperative period and the benefits and benefits of the patient's recovery process will be determined. Thus, effective application can be made for the entire postoperative period. It is thought that this study to be conducted will be a guide for future studies on the patient group.

DETAILED DESCRIPTION:
Intubation-based pharyngeal traumas are common in patients undergoing general anesthesia among the causes of post-operative sore throat and thirst symptoms. In the literature, it is reported that sore throat is frequently seen after endotracheal intubation (14.4% to 100%) and is one of the complications that patients fear most. Since sore throat and thirst can cause swallowing and breathing difficulties in the postoperative period, this affects the patient's nutrition and fluid intake and may prolong the recovery period. Also these are; creates a physical stress source, increases postoperative morbidity and reduces patient satisfaction. As pharmacological methods for relieving sore throat and thirst, it is recommended to use steroids and local anesthetics in the form of mouth washes and sprays. As non-pharmacological methods, it has been determined that aromatherapy, especially lavender, is effective in preventing and reducing sore throat and thirst. It has been determined that lavender has functions that reduce throat irritation, hoarseness, pain and stress among aromatic plants.

Postoperative nausea and vomiting (PONC) can be seen in 70-80% of surgical patients, and PONC, which is a side effect of anesthesia, is one of the most common complaints together with pain and thirsty. The American Society of Perianesthesia Nurses (ASPAN; American Society of PeriAnesthesia Nurses) defines POBK as nausea and vomiting seen within the first 24 hours after surgery. Aromatherapy is the most commonly used non-pharmacological alternative in the treatment of POBD. Ginger in aromatherapy applications; It is seen that it has been used effectively on gastrointestinal system diseases (gas remover, antispasmodic, appetite stimulant, aids in digestion and prevents nausea and vomiting) from ancient times all over the world.

Location and Features of the Research:

The study will be applied to individuals who have undergone percutaneous nephrolithotomy (PNL) in the urology clinic of Çukurova University Medical Faculty Balcalı Hospital. The urology clinic is a unit with a total of 36 patient beds, where emergency and elective surgeries are performed, and consists of 1 polyclinic and 1 department.

Universe and Sample:

The population of the study will be the patients who underwent PNL (percutaneous nephrolithotomy) operation in the urology clinic of Çukurova University Faculty of Medicine. The sample of the study will consist of patients who underwent PNL operation, met the inclusion criteria, and voluntarily agreed to participate in the study. The analgesic and antiemetic drugs that are routinely applied in the clinic after the surgery will continue, that is, the routine medical treatment of the patients will be carried out and will not be discontinued.

Data Collection Tools:

Prepared by the researcher in data collection; Informed consent form, personal information form, visual assessment scale (VAS - Visual Analog Scale) for the measurement of postoperative thirst and sore throat, and postoperative verbal descriptive scale (VDS - Verbal Descriptive Scale) will be used to evaluate nausea-vomiting. Statistical analysis of the collected data will be done using a package program called SPSS (IBM SPSS Statistics 24).

Ethical Permission:

Before starting the research, permission was obtained from Çukurova University Faculty of Medicine, Balcalı Hospital, Urology Department and Balcalı Hospital Chief Physician, dated 13.11.2020 and numbered E.137729. The permission of the Traditional and Complementary Medicine Clinical Research Ethics Committee, dated 13.01.2021 and numbered 23, was obtained.

The products to be used in the aromatic solution and the preparation dose rates, approved by the General Directorate of Health Services of the Ministry of Health, IU/Fito/01-03 for the year 2020, Gaziosmanpaşa University Anesthesiology and Reanimation Department Lecturer Prof. Dr. It was determined under the consultancy of Mustafa Süren. In addition, in the urology department where the research will be conducted, mouth spray application is routinely used in cases deemed appropriate for post-operative patients. Therefore, a study was planned to examine the effect of using these solutions during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Accepting the research
* Elective surgery planned with general anesthesia
* Patients in Asa I, II and III classes
* No hearing problem
* No history of allergies to lavender and ginger
* One-time intubation and no difficult intubation
* Those who have no previous psychiatric or mental illness will be included.

Exclusion Criteria:

* Did not accept the research
* In addition to clinical routine medical treatment, extra drug administration
* Patients with suspected aspiration risk will be excluded.

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-29 (Actual)

PRIMARY OUTCOMES:
Nonpharmacological method effects (Sore Throat) | postoperative first day
  Visual assessment scale (VAS) will be used to measure sore throat in the study. In this method, the person will be told that there are two endpoints from 1 to 10 that indicate whether they have a sore throat and that they should mark anywhere between these points.
  It is a scale evaluated by patients by making signs on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very well and the other end is indicating that the patient is very bad.
  VAS measurement will be performed 0, 2, 4, 6 and 8 hours after the patients are transferred from the anesthesia recovery unit to the clinic where they normally lie down after the surgery and are placed in their beds. The experiment will be applied to the placebo and control groups.
Nonpharmacological method effects (Thirst) | postoperative first day
  Visual assessment scale (VAS) will be used to measure thirst in the study. In this method, the person will be explained that there are two endpoints from 1 to 10 that indicate whether they have a sore throat and that they should mark anywhere between these points.
  It is a scale that is evaluated by the patients by making markings on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very good the other end is very bad.
  VAS measurement will be performed at 0, 2, 4, 6, and 8 hours after the patients are transferred from the anesthesia resting unit to the clinic where they are normally hospitalized after the surgery and are placed in their beds. The experiment will be applied to the placebo and control groups.
Nonpharmacological method effects (Nausea and Vomiting) | postoperative first day
  In the measurement of nausea-vomiting, a five-stage verbal descriptive scale (VDS) will be applied postoperatively (None: 0, mild nausea: 1, moderate nausea and vomiting: 2, frequent vomiting: 3, severe vomiting: 4).
  VDS will be measured at 0, 2, 4, 6 and 8 hours after the patients are transferred from the anesthesia resting unit to the clinic where they normally lie down after the surgery and are placed in their beds. The experiment will be applied to the placebo and control groups.

SECONDARY OUTCOMES:
Nonpharmacological method effects (Sore Throat) | postoperative first day
  Visual assessment scale (VAS) will be used to measure sore throat in the study. In this method, the person will be told that there are two endpoints from 1 to 10 that indicate whether they have a sore throat and that they should mark anywhere between these points.
  It is a scale evaluated by patients by making signs on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very well and the other end is indicating that the patient is very bad.
  VAS measurement will be performed 0, 2, 4, 6 and 8 hours after the patients are transferred from the anesthesia recovery unit to the clinic where they normally lie down after the surgery and are placed in their beds.
  It will be done after the aroma solution application to the experimental group. It will be done after the drinking water application to the placebo group. It will not be done because no intervention was applied to the control group.
Nonpharmacological method effects (Thirst) | postoperative first day
  Visual assessment scale (VAS) will be used to measure thirst in the study. In this method, the person will be explained that there are two endpoints from 1 to 10 that indicate whether they have a sore throat and that they should mark anywhere between these points.
  It is a scale that is evaluated by the patients by making markings on a 10 cm or 100 mm horizontal or vertical line (or horizontal line with numbers from 1 to 10), with one end indicating that the patient is very good the other end is very bad.
  VAS measurement will be performed at 0, 2, 4, 6, and 8 hours after the patients are transferred from the anesthesia resting unit to the clinic where they are normally hospitalized after the surgery and are placed in their beds.
  It will be done after the aroma solution application to the experimental group. It will be done after the drinking water application to the placebo group. It will not be done because no intervention was applied to the control group.
Nonpharmacological method effects (Nausea and Vomiting) | postoperative first day
  In the measurement of nausea-vomiting, a five-stage verbal descriptive scale (VDS) will be applied postoperatively (None: 0, mild nausea: 1, moderate nausea and vomiting: 2, frequent vomiting: 3, severe vomiting: 4).
  VDS will be measured at 0, 2, 4, 6 and 8 hours after the patients are transferred from the anesthesia resting unit to the clinic where they normally lie down after the surgery and are placed in their beds.
  It will be done after the aroma solution application to the experimental group. It will be done after the drinking water application to the placebo group. It will not be done because no intervention was applied to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Süren, Phd Prof, Principal Investigator — Gaziosmanpaşa University Department of Anesthesiology and Reanimation
Locations (1):
- Cukurova University, Sarıçam, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chinachoti T, Pojai S, Sooksri N, Rungjindamai C. Risk Factors of Post-operative Sore Throat and Hoarseness. J Med Assoc Thai. 2017 Apr;100(4):463-8. PMID 29911921
- [Background] Agarwal A, Gupta D, Yadav G, Goyal P, Singh PK, Singh U. An evaluation of the efficacy of licorice gargle for attenuating postoperative sore throat: a prospective, randomized, single-blind study. Anesth Analg. 2009 Jul;109(1):77-81. doi: 10.1213/ane.0b013e3181a6ad47. PMID 19535697
- [Background] Ahmed A, Abbasi S, Ghafoor HB, Ishaq M. Postoperative sore throat after elective surgical procedures. J Ayub Med Coll Abbottabad. 2007 Apr-Jun;19(2):12-4. PMID 18183710
- [Background] Shrestha S , Maharjan B , Karmacharya RM . Incidence and Associated Risk Factors of Postoperative Sore Throat in Tertiary Care Hospital. Kathmandu Univ Med J (KUMJ). 2017 Jan.-Mar.;15(57):10-13. PMID 29446355
- [Background] Lee JY, Sim WS, Kim ES, Lee SM, Kim DK, Na YR, Park D, Park HJ. Incidence and risk factors of postoperative sore throat after endotracheal intubation in Korean patients. J Int Med Res. 2017 Apr;45(2):744-752. doi: 10.1177/0300060516687227. Epub 2017 Feb 7. PMID 28173712
- [Background] Tazeh-Kand NF, Eslami B, Mohammadian K. Inhaled fluticasone propionate reduces postoperative sore throat, cough, and hoarseness. Anesth Analg. 2010 Oct;111(4):895-8. doi: 10.1213/ANE.0b013e3181c8a5a2. Epub 2010 Mar 17. PMID 20237046
- [Background] Soltani R, Soheilipour S, Hajhashemi V, Asghari G, Bagheri M, Molavi M. Evaluation of the effect of aromatherapy with lavender essential oil on post-tonsillectomy pain in pediatric patients: a randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2013 Sep;77(9):1579-81. doi: 10.1016/j.ijporl.2013.07.014. Epub 2013 Aug 8. PMID 23932834
- [Background] Smith HS, Smith EJ, Smith BR. Postoperative nausea and vomiting. Ann Palliat Med. 2012 Jul;1(2):94-102. doi: 10.3978/j.issn.2224-5820.2012.07.05. PMID 25841469
- [Background] American Society of PeriAnesthesia Nurses PONV/PDNV Strategic Work Team. ASPAN'S evidence-based clinical practice guideline for the prevention and/or management of PONV/PDNV. J Perianesth Nurs. 2006 Aug;21(4):230-50. doi: 10.1016/j.jopan.2006.06.003. No abstract available. PMID 16935735
- [Background] Oh KE, Song AR, Sok SR. Effects of Aroma Gargling, Cold Water Gargling, and Wet Gauze Application on Thirst, Halitosis, and Sore Throat of Patients After Spine Surgery. Holist Nurs Pract. 2017 Jul/Aug;31(4):253-259. doi: 10.1097/HNP.0000000000000219. PMID 28609410
- [Background] Sedigh Maroufi S, Moradimajd P, Moosavi SAA, Imani F, Samaee H, Oguz M. Dose Ginger Have Preventative Effects on PONV-Related Eye Surgery? A Clinical Trial. Anesth Pain Med. 2019 Oct 22;9(5):e92072. doi: 10.5812/aapm.92072. eCollection 2019 Oct. PMID 31903330
- [Background] Fearrington MA, Qualls BW, Carey MG. Essential Oils to Reduce Postoperative Nausea and Vomiting. J Perianesth Nurs. 2019 Oct;34(5):1047-1053. doi: 10.1016/j.jopan.2019.01.010. Epub 2019 May 27. PMID 31147268
- [Derived] Gokce E, Yurtseven S, Arslan S, Suren M, Akdogan N. The effect of an aromatic solution applied after percutaneous nephrolithotomy on sore throat, thirst, and nausea-vomiting: A randomised controlled trial. Complement Ther Clin Pract. 2025 Feb;58:101934. doi: 10.1016/j.ctcp.2024.101934. Epub 2024 Dec 6. PMID 39644858